CLINICAL TRIAL: NCT04602754
Title: National, Multicenter, Randomized, Double-blind, Triple-dummy, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Berlim 25/20 Association in the Treatment of Type II Diabetes Mellitus and Dyslipidemia.
Brief Title: Efficacy and Safety of Berlim 25/20 Association in the Treatment of Type II Diabetes Mellitus and Dyslipidemia.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS1019 - Berlim 25/20
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Dyslipidemia Associated With Type II Diabetes Mellitus
Keywords: Dyslipidemia; Type II Diabetes Mellitus
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2 | interventions — empagliflozin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BERLIM 25/20 (Experimental): The study is triple-dummy. The patient must take 3 tablets once a day, as follows:
  1 tablet Berlim 25/20 association, oral;
  1 tablet empagliflozin placebo, oral;
  1 tablet rosuvastatin calcium placebo, oral.
  Interventions: Drug: BERLIM 25/20 ASSOCIATION; Other: EMPAGLIFLOZIN PLACEBO; Other: ROSUVASTATIN CALCIUM PLACEBO
- Empagliflozin + rosuvastatin calcium (Active Comparator): The patient must take 3 tablets once a day, as follows:
  1 tablet Berlim 25/20 association placebo, oral;
  1 tablet empagliflozin, oral;
  1 tablet rosuvastatin calcium, oral.
  Interventions: Drug: EMPAGLIFLOZIN; Drug: ROSUVASTATIN CALCIUM; Other: BERLIM 25/20 ASSOCIATION PLACEBO

INTERVENTIONS:
Drug: BERLIM 25/20 ASSOCIATION — Berlim 25/20 association coated tablet.
  Arms: BERLIM 25/20
Other: EMPAGLIFLOZIN PLACEBO — Empagliflozin placebo coated tablet.
  Arms: BERLIM 25/20
Other: ROSUVASTATIN CALCIUM PLACEBO — Rosuvastatin calcium placebo coated tablet.
  Arms: BERLIM 25/20
Drug: EMPAGLIFLOZIN — Empagliflozin 25 mg coated tablet.
  Arms: Empagliflozin + rosuvastatin calcium
Drug: ROSUVASTATIN CALCIUM — Rosuvastatin 20 mg coated tablet.
  Arms: Empagliflozin + rosuvastatin calcium
Other: BERLIM 25/20 ASSOCIATION PLACEBO — Berlim 25/20 association placebo coated tablet.
  Arms: Empagliflozin + rosuvastatin calcium

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Berlim 25/20 association in the treatment of type 2 diabetes mellitus and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Participants of both sexes, with age greater than or equal to 18 years and less than or equal to 85 years;
* Participants presenting the diagnosis of type II diabetes mellitus, and who did not reach the therapeutic goals of HbA1c with previous dietary, physical exercise guidance and previous therapies at a stable dose in the last 3 months;
* HbA1c ≥ 7,5% and ≤ 10,5% and fasting blood glucose > 100 mg/dL at the screening visit;
* Participants with high or very high cardiovascular risk according to the Brazilian guideline on the prevention of cardiovascular diseases in patients with diabetes (2017), which have not reached the goal of LDL-c ≤ 70 mg/dL or ≤ 50 mg/dL, respectively, with lifestyle changes, who are or aren't using low or moderate potency statins;
* BMI (body mass index) > 19 Kg/m2 and ≤ 45 Kg/m2.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* History of alcohol abuse or illicit drug use;
* Participation in a clinical trial in the year prior to this study;
* Pregnancy or risk of pregnancy and lactating patients;
* Known hypersensitivity to the formula components used during the clinical trial;
* Type 1 diabetes mellitus;
* Fasting blood glucose > 300 mg/dL;
* Risk factors for volume depletion;
* Participants with total cholesterol > 500 mg/dL or triglycerides > 500 mg/dL;
* Impaired renal function and end-stage renal disease;
* Participants with known heart failure, class III to IV (New York Heart Association);
* Impaired hepatic function;
* Medical history of pancreatic diseases that may suggest insulin deficiency;
* Participants who had any cardiovascular event (acute myocardial infarction, acute coronary syndrome, recent onset stable angina, stroke, unstable congestive heart failure requiring treatment change), underwent revascularization or vascular surgery in the 6 months prior to screening;
* Bariatric surgery in the last two years and/ or other gastrointestinal surgeries that can cause chronic malabsorption syndrome;
* Condition that, in the investigator's judgment, may favor clinically significant changes in CPK levels;
* Current medical history of cancer and/ or cancer treatment in the last 5 years;
* Participants with known uncontrolled hypothyroidism or TSH levels > 5 mIU/L;
* History of known muscle disease or prior statin intolerance;
* Participants using SGLT2 inhibitors, sulfonylureas and/or insulin therapy or PCSK9 inhibitors;
* Participants who used other medications with prominent action in the control of serum triglyceride and cholesterol levels in the last 4 weeks or who are using low or moderate-intensity statins that cannot be replaced by rosuvastatin 20 mg;
* Participants using medications that may interfere with triglyceride and cholesterol metabolism started less than 4 weeks ago or with dose adjustment in the last 4 weeks prior to the screening visit;
* Treatment with anti-obesity drugs for less than 2 months or with dose change in the last 2 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of glycated hemoglobin levels measured between the first visit and the last visit. | 120 days
Percentual reduction of LDL-c levels measured between the first visit and the last visit. | 120 days

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 150 days

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa, Campinas, São Paulo, Brazil